CLINICAL TRIAL: NCT03965013
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneous NNC0268-0965 in Healthy Subjects and in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study to Look at How Safe NNC0268-0965 is in Healthy People and People With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1965-4456; 2018-003922-98 (Registry Identifier: European Medicines Agency (EudraCT)); U1111-1221-9696 (Registry Identifier: World Health Organization (WHO))
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 1; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts each with 2 arms. Part 1 is NNC0268-0965 vs. placebo in healthy volunteers. Part 2 is NNC0268-0965 vs. insulin glargine in subjects with type 1 diabetes mellitus.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 (healthy): NNC0268-0965 (Experimental): A single dose of NNC0268-0965 given s.c. (subcutaneously, under the skin)
  Interventions: Drug: NNC0268-0965
- Part 1 (healthy): placebo (Placebo Comparator): A single dose of placebo (NNC0268-0965) given s.c.
  Interventions: Drug: Placebo
- Part 2 (type 1 diabetes): NNC0268-0965 (Experimental): A single dose of NNC0268-0965 given s.c.
  Interventions: Drug: NNC0268-0965
- Part 2 (type 1 diabetes): insulin glargine (Active Comparator): A single dose of insulin glargine given s.c.
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: NNC0268-0965 — 2 to 3 dose levels will be tested in Part 1. 3 to 5 dose levels will be tested in Part 2
  Arms: Part 1 (healthy): NNC0268-0965; Part 2 (type 1 diabetes): NNC0268-0965
Drug: Placebo — A single dose of placebo given in Part 1
  Arms: Part 1 (healthy): placebo
Drug: insulin glargine — Insulin glargine given at a fixed dose level of 0.5 U/kg
  Arms: Part 2 (type 1 diabetes): insulin glargine

SUMMARY:
This study is investigating the safety and tolerability of the new medicine NNC0268-0965 (referred to as insulin 965), its concentrations in the blood and its effect on blood sugar for the treatment of diabetes. This first part of the study is conducted in healthy people, while there is a second part involving people with type 1 diabetes. The study will test how insulin 965 is tolerated by the participants' body, how it is taken up in the participants' blood, how long it stays there and how blood sugar is lowered. Participants will either get the new insulin 965 or placebo (an injection that does not contain active medicine) - which treatment you get is decided by chance. It is the first time that insulin 965 is tested in humans. Participants will get one injection of either insulin 965 or placebo under the skin of the left thigh. The study will last for about 5 weeks. Participants will have 6 clinic visits with the study doctor. People cannot be in the study if the study doctor thinks that there are risks for their health.

ELIGIBILITY:
Inclusion Criteria:

* Part 1 (healthy subjects):

  1. Male, aged 18-55 years (both inclusive) at the time of signing informed consent.
* Part 2 (subjects with type 1 diabetes mellitus):

  1. Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent.
  2. Diagnosed with type 1 diabetes mellitus equal to or more than1 year prior to the day of screening.
  3. Male subject or female subject of non-child bearing potential. Non-child bearing potential being surgically sterilized (i.e. documented hysterectomy, bilateral salpingectomy or bilateral oophorectomy or being postmenopausal (as defined as no menses for 12 months without an alternative medical cause).
  4. Current daily total insulin treatment between 0.2 (I)U/kg/day and 1.2 (I)U/kg/day (both inclusive).
  5. HbA1c equal to or below 8.5%.
  6. Fasting C-peptide below 0.30 nmol/L.

Exclusion Criteria:

* (Part 1 and Part 2) 1. Male of reproductive age who or whose partner(s) is not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice). Adequate contraceptive measures include that the male subject uses a condom during intercourse and that the partner practices adequate contraception (risk of pregnancy must be lower than 1%). In addition, subjects must not donate sperm for the duration of the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-12-14 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events | From trial product administration at day 1 until completion of post-treatment end-of-trial visit at day 10
  Number of events

SECONDARY OUTCOMES:
Number of treatment-emergent hypoglycaemic episodes | From trial product administration at day 1 until completion of post-treatment end-of-trial visit at day 10
  Number of episodes
Area under the serum NNC0268-0965 concentration-time curve after a single dose | From 0 hours until infinity after trial product administration (day 1)
  pmol*h/L
Maximum observed serum NNC0268-0965 concentration after a single dose | From 0 hours until last measurement time after trial product administration (day 1)
  pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com